CLINICAL TRIAL: NCT03662048
Title: Improving Infant Sleep Safety With the Electronic Health Record: Using Infant Photographs Taken by Parents for Individualized Feedback
Brief Title: Improving Infant Sleep Safety With the Electronic Health Record
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Milton S. Hershey Medical Center (Other)
Responsible Party: Principal Investigator, Ian M. Paul, MD, Professor of Pediatrics and Public Health Sciences Chief, Division of Academic General Pediatrics Vice Chair of Faculty Affairs, Department of Pediatrics, Milton S. Hershey Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: STUDY00010450
Record Dates: First submitted 2018-09-05; First posted 2018-09-07 (Actual); Last update posted 2019-10-11 (Actual); Status verified 2019-10

CONDITIONS: SIDS; Infant Development
MeSH Terms: conditions — Sudden Infant Death | interventions — Risk Evaluation and Mitigation

STUDY DESIGN:
Who Masked: Care Provider
Masking Description: 2 month photographs will be evaluated by study team members blinded to the study group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention at 1 month + usual care (Active Comparator): Parents will send the study team photographs of their infant sleeping during the night at ages 1 and 2 months.
  Interventions: Behavioral: Safe
- usual care (Placebo Comparator): Parents will send the study team photographs of their infant sleeping during the night only at at age 2 months.
  Interventions: Behavioral: Safe

INTERVENTIONS:
Behavioral: Safe — Feedback, according to the 2016 national American Academy of Pediatrics (AAP) guidelines on Sudden Unexplained Infant Death (SUID) risk factors, will be generated by the study team and communicated with parents. Feedback will be given to parents in the intervention group at ages 1 and 2 months. The control group parents will only receive this feedback at age 2 months.

SUMMARY:
This research is being done to find out if individualized feedback provided to parents on safe infant sleep can improve safety. This will be accomplished by having parents send photographs of their baby sleeping through the patient portal of the electronic health record (EHR).

DETAILED DESCRIPTION:
The purpose of this study is to assess if photographs of infants sleeping at night sent by parents through the patient portal of the electronic health record (EHR) can be used to a) deliver individualized feedback on safe infant sleep surfaces and sleep health and b) improve parental knowledge of and adherence to guidelines for safe infant sleep surfaces and sleep health. The feasibility of this approach will also be assessed through a randomized, clinical trial involving 130 infants with primary care through Penn State Health. Participants will be randomized to receive personalized feedback on the infant sleep position and surface at age 1 month in addition to usual care or a usual care group. Both groups will receive personalized feedback on the infant sleep position and surface at infant age 2 months.

ELIGIBILITY:
Inclusion Criteria:

* Gestational age: ≥37 weeks
* Singleton birth
* Newborns ages 0 days to 14 days old
* Newborn nursery stay <=7 days
* English speaking mother
* Mother ≥18 years old
* Has email/internet access
* Willing to sign up for the Penn State Health Patient Portal through the Electronic Health Record (EHR)
* Owns a smart phone, digital camera, or tablet that can take pictures to be transmitted through the EHR
* Plan to follow with a Penn State Health Provider though the infant's 3-4 month well child visit

Exclusion Criteria:

* Maternal morbidity or pre-existing condition that affects ability to care for the newborn (e.g. narcotic drug use, chemotherapy, uncontrolled depression etc.)
* Child is being adopted or will not be in the care of the mother

Max Age: 14 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 130 (Actual)
Dates: Start 2018-10-30 (Actual); Primary Completion 2019-09-11 (Actual); Study Completion 2019-09-11 (Actual)

PRIMARY OUTCOMES:
percentage of infants who do not meet all AAP recommendations for sleeping environments at age 2 months | 2 months of age
  Safe sleep environment will include:
  1. Solitary vs. non-solitary sleep
  2. Supine vs. non-supine infant sleep position
  3. No loose objects vs. loose objects on the sleep surface
  4. Tight-bedding vs. loose-bedding
  5. Firm vs. soft sleep surface (i.e. crib/bassinete vs. sofa/bouncy chair)
  6. Infant's sleeping in same room as parents vs. separate room
  7. No head coverings vs. head coverings

SECONDARY OUTCOMES:
Parent compliance | 1 and 2 months of age
  Proportion of parents that send photographs of their infant's sleep environment at ages 1 month (intervention group) and 2 months (both groups)

CONTACTS AND LOCATIONS:
Overall Officials: Ian M Paul, MD, MSc, Principal Investigator — Penn State Hershey Milton S Hershey Medical Center
Locations (1):
- Penn State Milton S Hershey Medical Center, Hershey, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No
no plan to IPD with other researchers

REFERENCES:
- [Background] TASK FORCE ON SUDDEN INFANT DEATH SYNDROME. SIDS and Other Sleep-Related Infant Deaths: Updated 2016 Recommendations for a Safe Infant Sleeping Environment. Pediatrics. 2016 Nov;138(5):e20162938. doi: 10.1542/peds.2016-2938. Epub 2016 Oct 24. PMID 27940804
- [Derived] Canty EA, Fogel BN, Batra EK, Schaefer EW, Beiler JS, Paul IM. Improving infant sleep safety via electronic health record communication: a randomized controlled trial. BMC Pediatr. 2020 Oct 8;20(1):468. doi: 10.1186/s12887-020-02369-2. PMID 33032546